CLINICAL TRIAL: NCT02145533
Title: Evaluation of Plasma and Tissue Levels of Metalloproteinases and Neutrophil Gelatinase-associated Lipocalin in Arterial Aneurysms.
Brief Title: Matrix Metalloproteinases (MMPs),Neutrophil Gelatinase-associated Lipocalin (NGAL) Tissue and Plasma Levels and Aneurysms
Status: Completed | Type: Observational
Sponsor: University of Catanzaro (Other)
Responsible Party: Principal Investigator, Luca Gallelli, MD, University of Catanzaro
Other Study IDs: SURVAS
Record Dates: First submitted 2014-05-19; First posted 2014-05-23 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: MMPs and NGAL in Ruptured and Non-ruptured Aneurysms
Keywords: MMP; NGAL; Arterial Aneurysms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Group I: patient with ruptured aneurysms
- Group II: patients with non-ruptured aneurysms
- Group III: Healthy volunteers

SUMMARY:
An association between arterial aneurysms and matrix metalloproteinases (MMPs) has been described previously. MMPs regulate extracellular structural proteins and tissue remodeling. Neutrophil Gelatinase-associated Lipocalin (NGAL) is involved in the regulation of MMP activity. The aim of this work was to study the relationship between the levels of MMPs and NGAL and arterial aneurysms.

In a multicenter, open label, parallel groups, prospective study, patients with aneurysmal disease were divided into two groups: Group I (with ruptured aneurysm) and Group II (with non-ruptured aneurysm). Healthy volunteer patients were also enrolled and represented the control group (Group III).

The investigators enrolled 307 patients (Group I: 107, Group II: 200) with arterial aneurysm: 49 popliteal, 31 common femoral, 2 superficial femoral, 29 common iliac artery, 3 common carotid and 193 abdominal aorta. Finally, 11 healthy volunteer patients (9 males and 2 females, age range 40-70 year-old, median 56) were enrolled in Group III.

Elisa test and Western blot analysis revealed greater levels of immunoreactive MMP-9 and NGAL in all patients with ruptured aneurysms, both central and peripheral aneurysms, and in the aneurismal vessels.

These results provide important advances in the understanding of the natural history of arterial aneurysms. MMPs and NGAL play a role in development of arterial aneurysms and they may represent molecular markers for the prevention of aneurysmal rupture

DETAILED DESCRIPTION:
In the present study, the analysis of MMPs levels in plasma and tissues in patients with aneurysmal lesions identified several patterns of protease activity. Levels of both MMP-9 and NGAL were increased in aneurismal vessels, while the patterns of MMP-9 and NGAL expression was very high in all patients with ruptured aneurysm, both central and peripheral. These results show: 1) the chronic and degenerative nature of the aneurysmal lesion which is associated with increased levels of inflammatory proteinases, like MMP-9; 2) the apparent pivotal role of MMP-9 and NGAL in the pathophysiologic processes which lead to the final stage of natural history of aneurysms; and 3) the ubiquitous distribution of MMP-9 and NGAL. The pattern increased expression of MMP-9 and NGAL appears to be specific for aneurysmal arteries and it is not dependent on the anatomic site of the lesion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the diagnosis of arterial aneurysmal disease

Exclusion Criteria:

* History of cancer
* Hepatic failure
* Infectious or autoimmune diseases
* Patients requiring endovascular treatment.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of aneurysmal disease (central and peripheral, ruptured and non-ruptured).
Sampling Method: Non-Probability Sample
Enrollment: 307 (Actual)
Dates: Start 2010-01; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of MMPs levels in ruptured and non-ruptured aneurysms | 52 months
  MMPs plasma levels are evaluated via ELISA test. MMPs tissue levels are evaluated via Immunoblotting using anti MMPs monoclonal antibodies
Evaluation of NGAL levels in ruptured and non-ruptured aneurysms | 52 months
  NGAL plasma levels are evaluated via ELISA test. NGAL tissue levels are evaluated via Immunoblotting using anti NGAL monoclonal antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Stefano de Franciscis, M.D., Study Chair — University Magna Graecia of Catanzaro; Raffaele Serra, Principal Investigator — University Magna Graecia of Catanzaro
Locations (1):
- University of Catanzaro, Catanzaro, Italy